CLINICAL TRIAL: NCT02929563
Title: Pediatric Intensive Care Ulcer Prophylaxis Pilot Trial
Acronym: PIC-UP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2173
Record Dates: First submitted 2016-10-03; First posted 2016-10-11 (Estimated); Last update posted 2020-09-02 (Actual); Status verified 2020-09

CONDITIONS: Gastrointestinal Hemorrhage
MeSH Terms: conditions — Gastrointestinal Hemorrhage | interventions — Pantoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pantoprazole (Experimental): pantoprazole 1 mg/kg (maximum 40 mg) IV once daily until the participants no longer need mechanical ventilation - to a maximum of 30 days or until Pediatric Intensive Care Unit (PICU) discharge.
  Interventions: Drug: Pantoprazole
- placebo (for pantoprazole) (Placebo Comparator): an equivalent volume of normal saline IV once daily until the participants no longer need mechanical ventilation - to a maximum of 30 days or until PICU discharge.
  Interventions: Drug: Placebo (for pantoprazole)

INTERVENTIONS:
Drug: Pantoprazole
  Arms: pantoprazole
Drug: Placebo (for pantoprazole)
  Arms: placebo (for pantoprazole)

SUMMARY:
This study tests the feasibility of a large study of stress ulcer prophylaxis in critically ill children. Children admitted to the Pediatric Intensive Care Unit who are expected to require mechanical ventilation for more than 48 hours will be randomized to intravenous pantoprazole 1 mg/kg or matching placebo once daily until they no longer need mechanical ventilation.

DETAILED DESCRIPTION:
Despite sparse pediatric data on the effectiveness of stress ulcer prophylaxis to prevent gastrointestinal (GI) bleeding, 60% of critically ill children receive these medications. This may have unintended consequences - increasing the risk of nosocomial infections - which may be more serious and common than bleeding these drugs are prescribed to prevent. A large randomized trial (RCT) is needed to assess the balance of these risks and benefits, to determine if a strategy of withholding stress ulcer prophylaxis in critically ill children is not inferior to a strategy of routine stress ulcer prophylaxis. RCTs in pediatric critical care are exceptionally challenging to complete; thus, a rigorous pilot RCT is crucial. The pilot may prevent pursuit of a trial that is ultimately not feasible - which is ethically and financially responsible. It is more likely that this carefully designed pilot trial will ensure that the larger trial we undertake is successful.

ELIGIBILITY:
Inclusion Criteria:

1. less than 18 years of age
2. >4 months of age
3. requires respiratory support in the form of invasive mechanical ventilation, non-invasive mechanical ventilation, or high-flow oxygen
4. the attending physician expects the child to require respiratory support for at least 2 more days

Exclusion Criteria:

1. histamine-2 receptor antagonist (H2RA) or proton pump inhibitor (PPI) use for >1 week in the past month
2. active GI bleeding Blood in the nasogastric (NG) tube or coffee-ground emesis suspected by the attending physician to be from the oropharynx is not an exclusion criterion.
3. documented severe reflux, active H. pylori infection, severe esophagitis, Zollinger Ellison syndrome, Barrett's esophagus, peptic ulcer bleeding within 8 weeks
4. are receiving methylprednisolone 15 mg/kg/day or more (or equivalent) Equivalent doses: methylprednisolone, prednisone or prednisolone 15 mg/kg/day; dexamethasone 3 mg/kg/day; hydrocortisone 60 mg/kg/day
5. are receiving mycophenolate (enteral), methotrexate, nelfinavir, atazanavir, saquinavir, posaconazole
6. chronic ventilation on usual pressure settings and rate
7. nocturnal or intermittent non-invasive ventilation only
8. are eating, nursing, or if chronically fed via feeding tube, receiving usual feeds
9. received more than 1 daily-dose equivalent of acid suppressive medication in the PICU
10. were previously enrolled in this trial
11. are currently enrolled in a potentially confounding trial
12. are known to be pregnant or breastfeeding
13. are known to be allergic to pantoprazole or any other ingredient in the product
14. are not expected to survive this PICU admission because of palliative care or limited life support

Ages: 4 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 116 (Actual)
Dates: Start 2017-01-09 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Effective screening | During admission to the Pediatric Intensive Care Unit (to maximum of 30 days)
  We will consider the trial feasible if >80% of eligible patients are approached for consent.
Timely enrollment | During admission to the Pediatric Intensive Care Unit (to maximum of 30 days)
  We will consider the trial feasible if >80% of participants receive their first dose of the assigned study drug within 1 day of becoming eligible.
Participant accrual | During admission to the Pediatric Intensive Care Unit (to maximum of 30 days)
  We will consider the trial feasible if the average monthly enrollment is 2 or more participants per centre.
Protocol adherence | During admission to the Pediatric Intensive Care Unit (to maximum of 30 days)
  We will consider the trial feasible if >90% of doses are administered according to the protocol.

SECONDARY OUTCOMES:
Clinically important bleeding | During admission to the Pediatric Intensive Care Unit (to maximum of 30 days)
  Overt bleeding from the GI tract (can be hematemesis, nasogastric blood, melena, hematochezia) associated with one of the following within 24 hours: a decrease in hemoglobin of >20 g/L, hypotension (a decrease in systolic blood pressure of >10 mmHg or the need for new or increased doses of vasoactive medications), tachycardia (an increase in heart rate of >20 beats per minute) or a red blood cell transfusion.
Nosocomial infections | During admission to the Pediatric Intensive Care Unit (to maximum of 30 days)
  Ventilator associated pneumonia and C Difficile associated diarrhea
Other gastrointestinal bleeding | During admission to the Pediatric Intensive Care Unit (to maximum of 30 days)
  Bleeding from the gastrointestinal tract that is not clinically important (using the above criteria).

CONTACTS AND LOCATIONS:
Overall Officials: Mark Duffett, PhD, Principal Investigator — McMaster University
Locations (7):
- Canada (7):
  - Alberta Children's Hospital, Calgary, Alberta
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital, Hamilton, Ontario
  - Children's Hospital - London Health Science Centre, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - CHU Sainte-Justine, Montreal, Quebec
  - Montreal Children's Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Duffett M, Choong K, Foster J, Gilfoyle E, Lacroix J, Pai N, Thabane L, Cook DJ; Canadian Critical Care Trials Group. Pediatric intensive care stress ulcer prevention (PIC-UP): a protocol for a pilot randomized trial. Pilot Feasibility Stud. 2017 May 19;3:26. doi: 10.1186/s40814-017-0142-y. eCollection 2017. PMID 28533916